CLINICAL TRIAL: NCT02117076
Title: Blinded, Randomized Study of Gabapentin (Neurontin®) and Gabapentin Enacarbil (Horizant™) in Restless Leg Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment unsuccessful due to overly restrictive inclusion/exclusion criteria.
Sponsor: Theresa Zesiewicz, MD (Other)
Responsible Party: Sponsor-Investigator, Theresa Zesiewicz, MD, Professor of Neurology, Director USf Ataxia Center, University of South Florida
Organization: University of South Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLS and Gabapentin or Horizant
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Restless Leg Syndrome
Keywords: Restless leg syndrome; RLS; gabapentin; gabapentin enacarbil; Neurontin; Horizant
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gabapentin immediate release (Active Comparator): Gabapentin IR is the immediate release form of the medication. Subjects randomized to gabapentin IR will be started out at a dose of 300mg per day, taken one hour before bedtime for the first week. Daily dose will be increased by 300 mg daily every 4 days until 1200 mg of gabapentin IR is reached or until a stable, tolerated dose of gabapentin IR that relieves symptoms has been maintained for 2 weeks (IRLS scores less than 15). Those patients who cannot tolerate gabapentin IR will be allowed to down titrate by one dose level (300 mg daily), before dropping out of the study.
  Interventions: Drug: Gabapentin immediate release
- gabapentin enacarbil extended release (Active Comparator): Horizant is the extended release form of gabapentin enacarbil. Subjects randomized to Horizant will take 600mg at 5 pm. After four days of stable dosing of Horizant, subjects in this study group will be evaluated by phone for changes in RLS symptoms and Patient Global Impression scale to determine if a dose increase is warranted. Subjects in this group may be titrated up to 1200 mg daily during the 2 week titration period.
  Interventions: Drug: Gabapentin enacarbil extended release

INTERVENTIONS:
Drug: Gabapentin immediate release — up to 1200 mg per day
  Other Names: Neurontin
  Arms: gabapentin immediate release
Drug: Gabapentin enacarbil extended release — up to 1200 mg per day
  Other Names: Horizant
  Arms: gabapentin enacarbil extended release

SUMMARY:
The study will compare the safety, effectiveness and tolerability of gabapentin (Neurontin) versus gabapentin enacarbil (Horizant) as treatment restless leg syndrome.

DETAILED DESCRIPTION:
The study will compare the safety, effectiveness and tolerability of gabapentin (Neurontin) versus gabapentin enacarbil (Horizant) as treatment restless leg syndrome. Subjects will be randomized to gabapentin (IR) or Horizant™ (ER). Dosing will be blinded to both patient and study team members. Once study medication dosing has been optimized, subjects will then remain on a stable dose for six weeks until study endpoint, after which subjects will be down-titrated off of study medications.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with a diagnosis of primary restless leg syndrome using the International Restless Legs Syndrome Study Group (IRLSSG) diagnostic criteria8.
2. RLS symptoms ≥ 15 nights of the month prior to study enrollment and for ≥ 4 of 7 consecutive nights in the week prior to study enrollment (if untreated).
3. Age 18 years to 80 years.
4. International Restless Legs Scale (IRLS) Total severity score of ≥ 15 (moderate to severe severity). 8
5. Had significant sleep disturbance on item 4 of IRLS.8
6. Women of child-bearing potential must use a reliable method of contraception.
7. Informed consent. Subject must be willing and able to complete all study procedures.

Exclusion Criteria:

1. Any illness that in the investigator's opinion preclude participation in this study.
2. Subjects with non-RLS-related sleep disorders (e.g., sleep apnea)
3. Subjects with neurological diseases or movement disorders other than RLS (e.g., diabetic neuropathy, Parkinson's disease, multiple sclerosis, dyskinesias, and dystonias)
4. Pregnancy or lactation.
5. Concurrent participation in another clinical study.
6. Dementia or other psychiatric illness that prevents the patient from giving informed consent (Mini-Mental State Examination scores less than 27).
7. Legal incapacity or limited legal capacity.
8. History of RLS symptom augmentation or early-morning rebound with previous dopamine-agonist treatment.
9. Clinically significant abnormalities in renal function. 3,8,10
10. Presence of severe cardiovascular or pulmonary disease, bronchial asthma, renal, hepatic or endocrine disease.
11. Concomitant treatment with drugs known to affect sleep/wake, RLS or periodic limb movements, including antidepressants. Subjects receiving treatment for RLS at screening will be required to discontinue and wash out for a minimum of 5 half-lives.
12. Body mass index greater than 34 kg/m2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
International Restless Leg Syndrome Rating Scale (IRLS) | 10 weeks
  The IRLS is a measure of severity of Restless Legs Syndrome. It includes 10 items, measured on a scale of 0-4. A score of 1-10 indicates mild severity, 11-20 indicates moderate severity, 21-30 is severe and 31-40 is very severe. Primary outcome is the difference in IRLS scores for each of the treatment regimens.
  from 0 to 4.

SECONDARY OUTCOMES:
Restless Leg Syndrome Quality of Life Scale (RLSQoL) | Baseline, day 35, day 54.
  The Restless Legs Syndrome Quality of Life questionnaire (RLSQoL) assesses the impact of RLS on daily life, emotional well-being, social life, and work life.

OTHER OUTCOMES:
Medical Outcomes Study (MOS) Sleep Scale | Baseline, day 35, day 54
  The MOS Sleep Scale consists of 12 individual items (4 sleep disturbance, 2 sleep adequacy, 1 quantity of sleep and optimal sleep, 3 somnolence, 1 snoring, and 1 shortness of breath) and takes 5 to 10 minutes to complete. Question 1 is scored on a scale of 1 to 5 ( 1 = 0-15 min to more than 60 min) and Questions 2 to 12 are scored on a scale of 1 to 6 (1 = all of the time to 6 = none of the time. The Sleep Disturbance Subscale score is derived from the scores to Questions 1, 3, 7, and 8 and ranges from 0 to 100, where higher scores indicate greater sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Zesiewicz, MD, FAAN, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States